CLINICAL TRIAL: NCT04550533
Title: DESIGN AND VALIDATION OF A SCALE TO EVALUATE THERAPEUTIC ADHERENCE IN PATIENTS WITH ANTINEOPLASTIC DRUGS
Brief Title: DESIGN OF A SCALE TO MEASURE COMPLIANCE WITH DRUG TREATMENT IN PATIENTS WITH ORAL CHEMOTHERAPY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Elsa López Pintor, Dr, Universidad Miguel Hernandez de Elche
Other Study IDs: 18/327
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Therapeutic Adherence — To measure adherence to treatment in oncohematological patients in treatment with oral anti-cancer drugs

SUMMARY:
Introduction: In recent years, there has been an increase in the use of oral chemotherapy, for its comfort and for allowing a higher quality of life. However, one of the main drawbacks is the lack of adherence to treatment with important clinical, social and economic consequences. In this scenario, the investigators did not have a questionnaire designed and validated to measure adherence in onco-hematological patients, a population that was erroneously considered very adherent.

The objective of the investigators is to build and validate a questionnaire to measure adherence to treatment in oncohematological patients in treatment with oral anti-cancer drugs.

Methods and analysis: An observational study to validate questionnaires will be carried out combining qualitative and quantitative research techniques. With the results of a systematic review of the literature and a qualitative study based on focus groups, a questionnaire will be designed to measure adherence in oncohematological patients in treatment with with oral anti-cancer drugs. The investigators will include patiens from two hospitals in the Valencian Community.

Discussion: It is essential to have a simple, reliable and validated instrument for measuring adherence in cancer patients undergoing treatment with oral antineoplastic agents. With this, lack of therapeutic compliance and its causes can be detected in order to establish interventions that improve it.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 in treatment with oral anti-cancer drugs (groups L01 and L02 according to the ATC drug classification), that come to the San Juan Hospital or Elda General Hospital to collect their medication, will be included.

Exclusion Criteria:

* Those patients with communication difficulties, and/or do not agree to take part in the study, will be excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 in treatment with oral anti-cancer drugs (groups L01 and L02 according to the ATC drug classification) who come to hospital to collect their medication,
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Measure of therapeutic adherence | At least 3 month after treatment
  To build and validate a questionnaire to measure adherence to treatment in oncohematological patients in treatment with oral antineoplastic drugs

SECONDARY OUTCOMES:
Barriers and difficulties in evaluating adherence | At least 3 month after treatment
  To understand the barriers and difficulties in evaluating adherence to treatment with oral antineoplastic drug in oncohematological patients through a bibliographic search and by carrying out discussion groups with professionals and patients.